CLINICAL TRIAL: NCT02759757
Title: Is Kinesio Taping Able to Influence the Electrical Activity of Muscles in Patients With Low Back Pain? A Controlled Randomized Trial
Brief Title: Is Kinesio Taping Able to Influence the Electrical Activity of Muscles in Patients With Low Back Pain?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leandro Pires (Other)
Responsible Party: Sponsor-Investigator, Leandro Pires, PT, masters student, Universidade Cidade de Sao Paulo
Organization: Universidade Cidade de Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pires1904
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Low Back Pain
Keywords: Kinesio Taping; Low back Pain; Electromyographic; EMG
MeSH Terms: conditions — Low Back Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio Taping (Experimental): Patients from this group will receive the kinesio Taping® Tex Gold tape according to the manufacturer's instructions. Kinesio Taping will be applied for the purpose of inhibiting the erector spinal muscle from the twelfth thoracic vertebrae (longissimus portion) up to the first sacral vertebrae with 10 to 15% tension (paper-OFF) in a "I" position bilaterally.
  Interventions: Other: Kinesio Taping
- Placebo (Placebo Comparator): Patient from this group will receive a 5cm-wide Micropore® tape from the twelfth thoracic vertebrae (longissimus portion) up to the first sacral vertebrae bilaterally.
  Interventions: Other: Placebo
- Control (No Intervention): Patients allocated will not receive any intervention.

INTERVENTIONS:
Other: Kinesio Taping — This is a tape that can be placed in different parts of the body using different shapes and tensions. In theory, this tape can change muscle activity.
  Other Names: Kinesiology tape; Kinesio tape; Kinesiotaping
  Arms: Kinesio Taping
Other: Placebo — A micropore tape will be used as placebo
  Arms: Placebo

SUMMARY:
Objectives: To test if the Kinesio Tex Gold ® is able to change the electromyographic signal of iliocostalis and longissimus muscles in patients with chronic nonspecific low back pain.

Study design: Three-arm, randomized controlled trial with a blinded assessor.

Location of study: Physical therapy Clinic of the Universidade Cidade de São Paulo (UNICID)

Patients: Sixty-three patients with chronic nonspecific low back pain.

Intervention: Patients allocated to the Kinesio Taping® group will receive the tape as described by the manufacturer's manual. The patients assigned to the placebo group will receive a Micropore tape and the control group will not receive any intervention. All groups will be assessed before and 30 minutes after intervention

Measures: The following outcomes will be measured: 1) Muscle activity and 2) pain intensity.

Limitations: Therapists will not be blinded.

DETAILED DESCRIPTION:
Patients who are seeking care for low back pain at the physiotherapy clinic from Universidade São Paulo will be invited to participate in the study and informed about the objectives of the study and evaluation procedures.

Patients who agree to participate will sign a consent form.

Patients will be assessed at baseline and immediately after the interventions.

Investigators will collect data with regards to personal and anthropometric data, as well as pain intensity (measured by a 0-10 numerical rating scale in all follow up points) and disability (measured by the 0-24 point Roland Morris Disability Questionnaire at baseline only).

Finally, muscle activation will be evaluated by surface electromyography and the maximum voluntary contraction of the trunk at 30 degrees position for a lumbar dynamometer that will be adjusted to the anthropometric profile of patients. The average and maximum values of muscular strength will be obtained by maximum voluntary contraction. The electromyography will capture the muscle activity in an integrated manner to electrogoniometers and will transmit the data via Bluetooth to a desktop with a MWX8 software (Biometrics) that will analyze the data. Before instrumentation patients will be instructed to perform the trunk extension movement the therapist's commands to become familiar with the equipment. Soon after will be held instrumentation (placement of electromyography electrodes and electrogoniometers and lumbar dynamometer) maximal voluntary contraction will be collected in trunk extension without Kinesio taping

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain (with a duration of at least 3 months), with or without leg pain.

Exclusion Criteria:

* patients who have used the Kinesio Taping previously
* any contraindications to the use of Kinesio Tex Gold®, such as allergy or severe skin problems.
* patients with nerve root compromise
* patients with fracture, tumor, inflammatory and/or infectious diseases
* patients with severe cardiorespiratory and/or metabolic diseases
* previous spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Median Force | thirty minutes after interventions
  Median force (a measure of muscle activity) will be collected using surface electromyography.
Root Mean Square | thirty minutes after interventions
  Root Mean Square (a measure of muscle activity) will be collected using surface electromyography.

SECONDARY OUTCOMES:
Pain Intensity | thirty minutes after interventions
  This outcome will be measured using a 0-10 numerical rating scale ranging from "no pain" to "worse possible pain".

OTHER OUTCOMES:
Disability | baseline only
  Disability will be measured with a 0-24 Roland Morris Disability Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo OP Costa, PhD, Principal Investigator — Universidade Cidade de São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pires LG, Padula RS, Junior MADL, Santos I, Almeida MO, Tomazoni SS, Costa LCM, Costa LOP. Can Kinesio Taping(R) influence the electromyographic signal intensity of trunk extensor muscles in patients with chronic low back pain? A randomized controlled trial. Braz J Phys Ther. 2020 Nov-Dec;24(6):539-549. doi: 10.1016/j.bjpt.2019.12.001. Epub 2019 Dec 15. PMID 31866161